CLINICAL TRIAL: NCT01175096
Title: A Phase Ib, Open-label Study to Evaluate RAD001 as Monotherapy Treatment in Chinese Patients With Advanced Pulmonary Neuroendocrine Tumor
Brief Title: Safety and Tolerability Profile of RAD001 Daily in Chinese Patients With Advanced Pulmonary Neuroendocrine Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Prof.Yi-Long Wu, Vice-director of GGH, Guangdong Lung Cancer Institute, Guangdong General Hospital & Guangdong Academy of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001KCN01
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-05

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor
Keywords: neuroendocrine tumors; carcinoid tumor; RAD001 (everolimus, Afinitor®)
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Active Comparator): 2 x 5 mg (=10 mg) RAD001 p.o., once daily, at the same time each day Dose level modifications/interruptions must follow guidelines. One treatment cycle consists of 28 days.
  Interventions: Drug: RAD001 (everolimus, Afinitor®)

INTERVENTIONS:
Drug: RAD001 (everolimus, Afinitor®) — RAD001 will be provided by Novartis to the study sites. RAD001 is formulated as tablets of 5 mg strength, blister-packed under aluminum foil in units of 30 tablets. The study site will dispense an adequate supply of RAD001 to the patient for self-administration at home.
  2 x 5 mg (=10 mg) RAD001 p.o., once daily, at the same time each day, One treatment cycle consists of 28 days.
  Other Names: RAD001; everolimus; Afinitor®

SUMMARY:
RAD001 continues to be investigated as an anticancer agent on new indications such as neuroendocrine tumors (incl. carcinoid), breast cancer, liver cancer, gastric cancer and lymphoma based on its potential to act:

* directly on the tumor cells by inhibiting tumor cell growth and proliferation
* indirectly by inhibiting angiogenesis leading to reduced tumor vascularity (via potent inhibition of tumor cell HIF-1 activity and VEGF production and VEGF-induced proliferation of endothelial cells)

A role for RAD001 in combination with Sandostatin LAR® Depot in the treatment of advanced carcinoid tumor is suggested by data on the regulatory role of mTOR in cell growth and protein translation and the finding that somatostatin-induced growth arrest is mediated in part by inhibition of the PI3K pathway (Charland, et al. 2001).

The present study is designed to collect safety/tolerability data and evidences for efficacy of RAD001 in the medically highly unmet indication of advanced pulmonary neuroendocrine tumor in Chinese patients.

DETAILED DESCRIPTION:
The purpose of this phase I b study is to characterize the safety, tolerability, and efficacy of 10 mg RAD001 administered orally on a continuous once-daily dosing regimen in the treatment of advanced pulmonary neuroendocrine tumor. The neuroendocrine tumors arising from bronchi and lung account for 30% of all carcinoid tumors, and there are a lot of well differentiated adenocarcinoma, squamous cancer and large cell lung cancer with significant neuroendocrine carcinoma characteristics who seems had a similarly prognosis with carcinoid tumor. There is no effective treatment available for advanced pulmonary NETs at this time.

The rationale for this study is based on both preclinical and clinical considerations. IGF-1 is a known autocrine regulator of CgA secretion and cell growth in human neuroendocrine tumor cells (von Wichert, et al. 2000; Wulbrand, et al. 2000; Van Gompel and Chen 2004). A role for RAD001 as monotherapy in carcinoid and pancreatic NET is suggested by the regulatory role of mTOR in cell growth, metabolism and protein translation (Fingar and Blenis 2004; Vignot, et al. 2005) and the Novartis observation that the PI3K/mTOR pathway is activated by IGF-1 in carcinoid and pancreatic NET cells (von Wichert, et al. 2000; Van Gompel and Chen 2004).

The proposed RAD001 dosage regimen is 10 mg/day in both monotherapy and combination therapy settings. This regimen is based both on Novartis Phase I/II studies and on results from an investigator-sponsored study in NET. Initial Phase I studies of the RAD001 10 mg/day schedule demonstrated dose limiting toxicities in 2 of 12 patients. Tolerability of this schedule was verified in a total of 33 patients in Phase 1 studies as well as in 12 breast cancer patients treated with letrozole 2.5 mg plus RAD001 10 mg/day. Pharmacodynamic modeling indicates that downstream effectors of mTOR are completely suppressed by RAD001 at the 10 mg/day dose. No increased toxicity is expected from use of RAD001 in combination with Sandostatin LAR® Depot. The investigator-sponsored study in NET, toxicity observed with RAD001 5 mg/day in combination with Sandostatin LAR® Depot was similar to that observed for RAD001 5 mg/day alone in Phase 1 studies (Yao, et al. 2006). Therefore a dose of RAD001 10 mg/day will be evaluated in this study.

ELIGIBILITY:
For carcinoid tumor

Inclusion Criteria:

* Histologically confirmed carcinoid tumors
* Newly diagnosed advanced carcinoid tumors
* Measurable tumors
* Chinese men and women, age ≥ 18 years
* ECOG performance status ≤ 2
* Written informed consent obtained

Exclusion Criteria:

* Patients with either clinically apparent central nervous system metastases or carcinomatous meningitis(non-clinical symptoms with brain lesions is eligible)
* Received Cytotoxic chemotherapy, immunotherapy or radiotherapy prior to enrollment
* Patients with a concurrent malignancy, or history of prior malignancy within the past three years, except for basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, treated early stage (T1a) prostate cancer or treated early stage (DCIS or LCIS) breast cancer
* Prior therapy with RAD001 or other mTOR inhibitors (sirolimus, temsirolimus, everolimus)
* Major surgery in the past two weeks
* Any medical condition resulting in >CTC grade 2 dyspnea
* Patients with recent hemoptysis associated with carcinoid tumor (> 1 teaspoon in a single episode within 4 weeks)
* Serious, severe or uncontrolled medical or psychiatric condition
* Patients receiving chronic treatment with corticosteroids or another immunosuppressive agent
* Patients with a known history of HIV seropositivity
* Women of childbearing potential must have had a negative serum pregnancy test within 3 days prior to the administration of RAD001
* Patients who have received an investigative drug or therapy within the last 30 days

For adenocarcinoma and Large cell lung cancer with significant neuroendocrine carcinoma characteristics

Inclusion Criteria:

* Histologically confirmed locally unresectable or advanced well differentiated （adenocarcinoma,squamous cancer and large cell lung cancer ）with significant neuroendocrine carcinoma characteristics tumors : CgA and/or Synaptophysin +(at least 10% of cells that would have to be positive ).( the pathology shows a neuroendocrine component histologically should be at least 10% of tissue within the specimen that is read as "neuroendocrine component").
* Measurable tumors
* Patients with newly diagnosed advanced cancer or progressed after 1st line treatment is eligible
* Chinese men and women, age ≥ 18 years
* ECOG performance status ≤ 2
* Written informed consent obtained

Exclusion Criteria:

* Patients with either clinically apparent central nervous system metastases or carcinomatous meningitis(non-clinical symptoms with brain lesions is eligible)
* Radiotherapy to primary tumor in lung lesions prior to enrollment
* Patients with a concurrent malignancy, or history of prior malignancy within the past three years, except for basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, treated early stage (T1a) prostate cancer or treated early stage (DCIS or LCIS) breast cancer
* Prior therapy with RAD001 or other mTOR inhibitors (sirolimus, temsirolimus, everolimus)
* Major surgery in the past two weeks
* Any medical condition resulting in > CTC grade 2 dyspnea
* Patients with recent hemoptysis associated with carcinoid tumor (> 1 teaspoon in a single episode within 4 weeks)
* Serious, severe or uncontrolled medical or psychiatric condition
* Patients receiving chronic treatment with corticosteroids or another immunosuppressive agent
* Patients with a known history of HIV seropositivity
* Women of childbearing potential must have had a negative serum pregnancy test within 3 days prior to the administration of RAD001
* Patients who have received an investigative drug or therapy within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 28 ±4 days
  Safety assessments will consist of monitoring and recording all adverse events, including serious adverse events, the regular monitoring of hematology and blood chemistry, regular monitoring of vital signs and physical condition. A safety visit will take place on day 28 (±4 days) following the last dose of study drug administered. Patients will be asked to visit the clinic on day 1 of every 6 weeks for safety assessments. Safety and tolerability will be assessed according to the NIH/NCI CTC

SECONDARY OUTCOMES:
Tumor response | 6-week
  Tumor response will be evaluated at the end of every 6-week treatment period, Treatment will continue until tumor progression as judged by the local investigator using the RECIST criteria, unacceptable toxicity, death, or discontinuation from the study for any other reason.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD.PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital & Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China